CLINICAL TRIAL: NCT07273162
Title: The Effect of Cold Vapor Inhalation on Dyspnea Thirst Nausea and Physiological Parameters in the Recovery Unit After Laparoscopic Inguinal Hernia Surgery
Brief Title: The Effect of Cold Vapor on Dyspnea, Thirst, Nausea, and Physiological Parameters in the PACU After Laparoscopic Inguinal Hernia Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Yeliz Sürme, Assoc. Prof. Dr., TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2025-10/14
Record Dates: First submitted 2025-11-27; First posted 2025-12-09 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Patients Undergoing Laparoscopic Inguinal Hernia Repair
Keywords: PACU; Laparoscopy; inguinal hernia; cold vapor; dyspnea; thirst; nausea; physiological parameters; surgery
MeSH Terms: conditions — Hernia, Inguinal; Dyspnea; Nausea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: No information regarding group allocations will be shared with the expert statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold Vapor (Experimental): Immediately following the initial (T0) assessment of patients, in addition to routine care and treatment procedures, patients will receive cold vapor using the Hikoneb 906 S/LCD ultrasonic hospital-grade nebulizer device for 15 minutes. Following completion of the intervention, patients' status will be reassessed at 15 (T1) and 30 (T2) minutes.
  Interventions: Other: Cold Vapor
- Control Group (No Intervention): Patients in the control group will not be subjected to any additional intervention. Follow-up of patients in this group will be conducted in accordance with the clinic's current standard postoperative treatment and care practices, and patients will be evaluated at baseline (T0), 15 minutes (T1), and 30 minutes.

INTERVENTIONS:
Other: Cold Vapor — Cold steam application will be performed using a Hikoneb 906 S/LCD ultrasonic nebulizer, which will generate cold steam with distilled water. Device parameters will be optimally set to steam delivery level 5 (1-10), steam density level 5 (1-10), and steam temperature 1C0 (1C0-10C0). This application will be applied to the intervention group for 15 minutes after the baseline (T0) assessment. Cold steam will not be delivered directly to the airways but will be applied to the facial area, covering the mouth and nose area. A distance of approximately 20-30 cm will be maintained between the device's steam outlet and the patient's face.
  Arms: Cold Vapor

SUMMARY:
Cold vapor application is considered a promising intervention with the potential to alleviate side effects associated with anesthesia and surgery in the postoperative period. This study aims to determine the effect of cold vapor inhalation on dyspnea, thirst, nausea, and physiological parameters following laparoscopic inguinal hernia surgery.

Hypotheses (H1);

H1a: Patients administered cold vapor will report lower dyspnea severity compared to the control group.

H1b: Patients administered cold vapor will report lower thirst levels compared to the control group.

H1c: Patients administered cold vapor will report lower nausea severity compared to the control group.

H1d: Patients administered cold vapor will show significant differences in physiological parameters compared to the control group.

DETAILED DESCRIPTION:
Non-pharmacological methods, such as cold vapor application, hold significant potential in the management of complications encountered in the postoperative period. Despite this potential, to the best of our knowledge, no published study examining the effect of cold vapor on dyspnea, thirst, and physiological parameters has been found in the literature. This study is a randomized controlled experimental study. The study will be conducted with at least 66 patients in total, including 33 in the intervention group and 33 in the control group. Data collection consists of three stages: T0, T1, and T2. In these stages, the baseline (T0) assessment of both groups will be performed using the Questionnaire Form, Modified Borg Scale (MBS), Perioperative Thirst Discomfort Scale (PTDS), Numerical Rating Scale (NRS), and Physiological Parameter Follow-up Form (PPFF). Following this assessment, the patients' condition will be re-evaluated at the 15th minute (T1) and 30th minute (T2) using the MBS, PTDS, NRS, and PPFF. In the intervention group, immediately after the baseline (T0) assessment, cold steam application will be administered to patients for 15 minutes using a Hikoneb 906 S/LCD ultrasonic hospital-type nebulizer device, in addition to routine care and treatment procedures. Patients in the control group will not be subjected to any additional intervention. It is predicted that cold vapor inhalation will reduce the severity of dyspnea, thirst, and nausea after laparoscopic inguinal hernia surgery as a result of the study. Additionally, it is expected to bring basic vital parameter values such as systolic and diastolic blood pressure, heart rate (pulse/min), peripheral oxygen saturation (SpO2, %), and respiratory rate (/min) closer to the normal physiological range. This study is significant as it demonstrates the value of cold vapor as a practice that strengthens and supports individualized nursing care in the early postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being aged 18 years or older
* Being able to speak and understand Turkish
* Having cognitive, affective, and communicative competence
* Having intact visual and auditory functions
* Having undergone elective laparoscopic inguinal hernia surgery under general anesthesia
* Having an ASA score of I or II
* Having a total Modified Aldrete Score of ≥9 and a consciousness score of 2 (fully awake) in the postoperative period
* Not having developed vomiting prior to the intervention
* Having a body temperature within the normal physiological range (36-37.5 °C)

Exclusion Criteria:

* Having cold vapor application planned by physician order in the PACU prior to the study
* Having signs and symptoms of upper or lower airway obstruction
* Developing agitation and having communication insufficiency
* Having an allergy to cold vapor application
* Having a diagnosis of obstructive pulmonary disease (e.g., COPD, asthma) or heart failure
* Having a known history of any neurological or psychiatric disease
* Having a postoperative nasogastric catheter inserted
* Having received preoperative diagnoses associated with nausea, vomiting, or dyspnea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Survey Form | Baseline (T0)
  The form developed by the researchers consists of a total of 13 questions and collects data on the demographic (age (year), gender, body mass index (kg/m² ), ect.) and clinical characteristics (American Society of Anesthesiologists-ASA score, perioperative fasting period (min), ect.) of the patients.
Modified Borg Scale (MBS) for Dyspnea | Baseline (T0), 15th minute (T1) and 30th minute (T2)
  The MBS is a 12-point scale that rates dyspnea severity from 0 (no dyspnea) to 10 (intolerable dyspnea).
Numerical Rating Scale (NRS) for Nausea Level | Baseline (T0), 15th minute (T1) and 30th minute (T2)
  The severity of postoperative nausea in patients will be assessed using the NRS, which is scored from 0 to 10 and created by researchers. Higher scores on this scale represent higher severity of nausea.
Surgical Period Thirst-Related Discomfort Scale (SPTRDS) | Baseline (T0), 15th minute (T1) and 30th minute (T2)
  This six-item, three-point Likert-type scale has a single-dimensional structure. Items were rated as "did not bother" (0), "slightly bothered" (1), and "very bothered" (2). Higher scores on this scale represent higher severity of thirst.
Physiological Parameter Monitoring Form (PPMF) | Baseline (T0), 15th minute (T1) and 30th minute (T2)
  The monitoring form, created by the researcher as part of the study, will assess basic vital signs such as systolic (mmhg) and diastolic (mmhg) blood pressure, heart rate (pulse/min), peripheral oxygen saturation (SpO2, %) and respiratory rate (/min).

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No